CLINICAL TRIAL: NCT00568958
Title: Naltrexone for Heavy Drinking in Young Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0706002743; R01AA016621 (NIH); NIH grant AA016621-01
Record Dates: First submitted 2007-12-04; First posted 2007-12-06 (Estimated); Results first posted 2014-08-11 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2018-08

CONDITIONS: Alcohol Consumption; Alcoholic Intoxication; Alcoholism; Alcohol-induced Disorders
Keywords: heavy episodic drinking; young adults; naltrexone; BASICS counseling; alcohol-related consequences; double-blind trial; randomized clinical trial
MeSH Terms: conditions — Alcohol Drinking; Alcoholic Intoxication; Alcoholism; Alcohol-Induced Disorders | interventions — Crisis Intervention; Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Naltrexone (Experimental): Active naltrexone (25 mg daily +25 targeted)+ BASICS counseling
  Interventions: Behavioral: BASICS counseling; Drug: naltrexone
- Placebo Naltrexone (Placebo Comparator): Placebo Naltrexone (targeted + daily) + BASICS Counseling
  Interventions: Behavioral: BASICS counseling; Drug: placebo naltrexone

INTERVENTIONS:
Behavioral: BASICS counseling — Brief Alcohol Screening and Intervention for College Students (BASICS) is a form of counseling that was developed originally for use with undergraduates. It combines three main elements: motivational enhancement strategies, skills for moderating consumption, and provision of individualized feedback.
  Other Names: brief counseling; brief intervention
Drug: naltrexone — Daily + targeted (i.e., taken as needed in anticipation of a high-risk situation) naltrexone, 25mg each for a total possible dose of 50mg (the FDA-approved dose for alcohol dependence) in a given day for a period of 8 weeks.
  Other Names: ReVia; Depade
  Arms: Naltrexone
Drug: placebo naltrexone — Daily + targeted (i.e., taken as needed in anticipation of a high-risk situation) placebo for a period of 8 weeks.
  Arms: Placebo Naltrexone

SUMMARY:
In this study, 140 heavy drinking young adults (aged 18-25) will be provided with brief counseling and either naltrexone, a medication that is FDA-approved for the treatment of alcohol dependence, or placebo over the course of 8 weeks. A novel strategy will be used for administering low-dose naltrexone, in which daily dosing will be combined with targeted dosing in anticipation of high-risk situations. The main hypotheses are that daily + targeted naltrexone will result in greater reductions in frequency of heavy and any drinking compared with daily + targeted placebo.

DETAILED DESCRIPTION:
NIAAA has designated underage drinking as a priority research area. Of note, the highest prevalence of problem alcohol use is among young adults ages 18-25. Heavy drinking that occurs during this period can have important immediate and lifelong adverse consequences. Behavioral interventions, notably BASICS (Brief Alcohol Screening and Intervention for College Students), have been developed to help young adults reduce their drinking. Although these interventions are effective, including with college students mandated to treatment and others with minimal motivation to stop drinking, the effect sizes are modest, suggesting that new approaches are needed to enhance these interventions. A promising strategy yet to be tested in young adults is the use of the opiate antagonist naltrexone. In other research, naltrexone has been shown to reduce the amount of alcohol consumed, even in the absence of strong internal motivation to change, and to reduce the frequency of any and heavy drinking in problem drinkers seeking treatment. Thus we propose to conduct an 8 week double-blind placebo-controlled trial to test the combined efficacy of BASICS + naltrexone in 132 young adults aged 18-25 who drink heavily. A novel strategy will be used for administering low-dose naltrexone, in which daily dosing will be combined with targeted dosing in anticipation of high-risk situations. The main hypotheses are that daily + targeted naltrexone will result in greater reductions in frequency of heavy and any drinking compared with daily + targeted placebo. In order to enhance the sensitivity with which we are able to assess naltrexone's effects on drinking, daily ratings will be obtained during treatment. These will permit us to examine alternative measures of alcohol involvement (e.g., reports of subjective intoxication, estimated blood alcohol levels) in addition to the traditional measures based on number of drinks consumed. These data will also be used to examine potential mediators (e.g., craving, subjective effects of alcohol) of treatment response in order to better understand the effects of naltrexone. The durability of treatment effects will be examined at 3, 6 and 12 months after randomization. Demonstration of the efficacy of naltrexone in this population will provide the essential information needed for its adoption by college counseling centers and other health care settings committed to reducing the risk of heavy drinking in young adults.

ELIGIBILITY:
Inclusion Criteria:

Each subject must:

1. Be between the ages of 18 and 25;
2. Report heavy drinking 4 or more times in the past 4 weeks. Heavy drinking is defined as 4 or more drinks for women and 5 or more drinks for men on an occasion;
3. Be able to read English and show no evidence of significant cognitive impairment.
4. That women of child-bearing potential (i.e., who has not had a hysterectomy, bilateral oophorectomy, or tubal ligation), be nonlactating, practicing a reliable method of birth control, and have a negative urine pregnancy test prior to initiation of treatment.

Exclusion Criteria:

No subject may:

1. Exhibit current, clinically significant physical disease or abnormality on the basis of medical history, physical examination, or routine laboratory evaluation, including AST or ALT levels greater than 3 times normal or bilirubin levels greater than 110% of normal. Individuals with common medical conditions (e.g., asthma, diabetes mellitus, thyroid disease) that are adequately controlled and who have a relationship with a primary-care practitioner will not be excluded;
2. Exhibit serious psychiatric illness (i.e., schizophrenia, bipolar disorder, severe major depression, panic disorder, borderline personality disorder, organic mood or mental disorders, or substantial suicide or violence risk) by history or psychological examination;
3. Have a current diagnosis of DSM-IV drug dependence other than nicotine, or a lifetime history of DSM-IV opiate dependence;
4. Have a current DSM-IV diagnosis of alcohol dependence that is clinically severe defined by a) a history of seizures, delirium, or hallucinations during alcohol withdrawal, b) a Clinical Institute Withdrawal Assessment scale (Sullivan et al., 1989) score of > 8, c) report drinking to avoid withdrawal symptoms, or d) have had prior treatment of withdrawal.
5. Have used opioids or concomitant therapy with any psychotropic drug in the past month, except that subjects who are on a stable dose of a Selective Serotonin Reuptake Inhibitor for at least two months for the indications of Major Depressive Disorder, Premenstrual Syndrome (PMS), or Premenstrual Dysphoric Disorder (PMDD) will not be excluded; SSRIs are allowed due to their safety profile relative to other classes of antidepressants.
6. Have a history of hypersensitivity to naltrexone;
7. Be considered by the investigators to be an unsuitable candidate for receipt of an investigational drug.
8. The investigators may exclude participants who complete daily questionnaires on less than half of the days between intake and treatment.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2008-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie O'Malley, PhD, Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center - Substance Abuse Treatment Unit, New Haven, Connecticut, United States

REFERENCES:
- [Derived] O'Malley SS, Corbin WR, Leeman RF, DeMartini KS, Fucito LM, Ikomi J, Romano DM, Wu R, Toll BA, Sher KJ, Gueorguieva R, Kranzler HR. Reduction of alcohol drinking in young adults by naltrexone: a double-blind, placebo-controlled, randomized clinical trial of efficacy and safety. J Clin Psychiatry. 2015 Feb;76(2):e207-13. doi: 10.4088/JCP.13m08934. PMID 25742208

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred primarily through Facebook advertisements and fliers. Following initial screening by phone or online surveys, individuals were invited for intake conducted by the research assistant at an outpatient university research clinic where written informed consent was obtained.
Period: Allocation
Arm/Group | Naltrexone | Placebo Naltrexone
Started | 70 | 70
Completed | 61 | 67
Not Completed | 9 | 3
Not completed — Withdrawal by Subject | 7 | 3
Not completed — Physician Decision | 2 | 0
Period: Follow-Up
Arm/Group | Naltrexone | Placebo Naltrexone
Started | 61 | 67
Completed | 52 | 60
Not Completed | 9 | 7
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Physician Decision | 1 | 1
Not completed — Family Emergency | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naltrexone | Placebo Naltrexone | Total
Number analyzed (Participants) | 61 | 67 | 128
Age, Customized [Number; unit: participants]
  18-25 year olds | 61 | 67 | 128
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 22 | 40
  Male | 43 | 45 | 88
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 49 | 50 | 99
  Non-Caucasian | 12 | 17 | 29
Alcohol Use Diagnosis [Number; unit: participants]
  No Diagnosis | 16 | 11 | 27
  Alcohol Abuse | 11 | 14 | 25
  Alcohol Dependence | 34 | 42 | 76

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Heavy Episodic Drinking
Description: Self-reported drinking was primarily obtained through diary data, with the Timeline Follow-Back Interview (TLFB) used to replace missing data at baseline and at each biweekly visit over the 8-weeks.The eight weeks follow-up measure is summarized across all biweekly visits. Frequency of heavy episodic drinking is measured as 5 or more drinks in a day for males, and 4 or more drinks in a day for females. A standard drink was equivalent to 0.6 gm of absolute alcohol (e.g., 12-oz beer, 5-oz wine, or 1.5-oz, 80-proof liquor). Baseline measures captured the prior 4 weeks.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: percentage of heavy drinking days
Arm/Group | Naltrexone | Placebo Naltrexone
Number analyzed (Participants) | 61 | 67
percentage of heavy drinking days | 34.3 (16.76) | 33.4 (13.68)

2. Secondary Outcome: Number of Drinks Per Drinking Day
Description: Self-reported drinking was primarily obtained through diary data, with the Timeline Follow-Back Interview (TLFB) used to replace missing data at baseline and at each biweekly visit over the 8-weeks.The eight weeks follow-up measure is summarized across all biweekly visits. Baseline measures captured the prior 4 weeks.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: drinks per drinking day
Arm/Group | Naltrexone | Placebo Naltrexone
Number analyzed (Participants) | 61 | 67
drinks per drinking day | 6.7 (2.9) | 6.77 (5.9)

3. Primary Outcome: Frequency of Heavy Episodic Drinking
Description: Self-reported drinking was primarily obtained through diary data, with the Timeline Follow-Back Interview (TLFB) used to replace missing data at baseline and at each biweekly visit over the 8-weeks.The eight weeks follow-up measure is summarized across all biweekly visits.
  Frequency of heavy episodic drinking is measured as 5 or more drinks in a day for males, and 4 or more drinks in a day for females over an eight week period. A standard drink was equivalent to 0.6 gm of absolute alcohol (e.g., 12-oz beer, 5-oz wine, or 1.5-oz, 80-proof liquor).
Time Frame: eight weeks
Measure: Mean (Standard Deviation); unit: percentage of heavy drinking days
Arm/Group | Naltrexone | Placebo Naltrexone
Number analyzed (Participants) | 61 | 67
percentage of heavy drinking days | 21.6 (16.05) | 22.9 (13.20)

4. Secondary Outcome: Number of Drinks Per Drinking Day
Description: Self-reported drinking was primarily obtained through diary data, with the Timeline Follow-Back Interview (TLFB) used to replace missing data at baseline and at each biweekly visit over the 8-weeks.The eight weeks follow-up measure is summarized across all biweekly visits.
Time Frame: 8 Weeks
Measure: Mean (Standard Deviation); unit: drinks per drinking day
Arm/Group | Naltrexone | Placebo Naltrexone
Number analyzed (Participants) | 61 | 67
drinks per drinking day | 4.9 (2.28) | 5.9 (2.51)

5. Secondary Outcome: Percentage of Drinking to an Estimated Blood Alcohol Concentration (BAC) of .08 or Higher
Description: Self-reported drinking was primarily obtained through diary data, with the Timeline Follow-Back Interview (TLFB) used to replace missing data at baseline and at each biweekly visit over the 8-weeks.The eight weeks follow-up measure is summarized across all biweekly visits.
  BAL (Blood Alcohol Level) was estimated using data from the daily diaries based on the number of drinks consumed, the duration of drinking, and total body water (based on gender, age, height and weight) using Curtin's formula.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Naltrexone | Placebo Naltrexone
Number analyzed (Participants) | 61 | 67
percentage of days | 35.4 (28.40) | 45.7 (26.80)

6. Primary Outcome: Percent Days Abstinent From Drinking
Description: as for outcome 2
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: % days abstinent
Arm/Group | Naltrexone | Placebo Naltrexone
Number analyzed (Participants) | 61 | 67
% days abstinent | 43.3 (21.77) | 49.5 (14.69)

7. Primary Outcome: Percent Days Abstinent From Drinking
Description: as for outcome 4
Time Frame: 8 Weeks
Measure: Mean (Standard Deviation); unit: % days abstinent
Arm/Group | Naltrexone | Placebo Naltrexone
Number analyzed (Participants) | 61 | 67
% days abstinent | 56.6 (22.52) | 62.5 (15.75)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the 8 week treatment period between March 2008 and January 2012.
Arm/Group | Naltrexone | Placebo Naltrexone
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/67
Other Adverse Events (participants affected / at risk) | 52/61 | 46/67
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Naltrexone (N=61) | Placebo Naltrexone (N=67)
Rash (Skin and subcutaneous tissue disorders) | 9 | 6
Itching (Skin and subcutaneous tissue disorders) | 8 | 5
Sweating (Skin and subcutaneous tissue disorders) | 4 | 2
Nausea (Gastrointestinal disorders) | 22 | 16
Vomiting (Gastrointestinal disorders) | 14 | 11
diarrhea (Gastrointestinal disorders) | 4 | 7
Abdominal Pain (Gastrointestinal disorders) | 4 | 6
Fatigue (General disorders) | 11 | 6
Decreased Appetite (General disorders) | 7 | 9
Increased Appetite (General disorders) | 5 | 7
Headache (Nervous system disorders) | 31 | 23
Insomnia (Nervous system disorders) | 12 | 14
Dizziness (Nervous system disorders) | 8 | 7
Sleepiness (Nervous system disorders) | 10 | 2
Anxiety (Psychiatric disorders) | 18 | 14
Depression (Psychiatric disorders) | 4 | 7
Irregular Menses (Reproductive system and breast disorders) | 4/18 | 4/22
Change in Libido (Reproductive system and breast disorders) | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No